CLINICAL TRIAL: NCT03050333
Title: Efficacy and Safety of Endoscopic Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EDUARDO ALBENIZ (Other)
Collaborators: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor-Investigator, EDUARDO ALBENIZ, MD, Fundacion Miguel Servet
Organization: Fundacion Miguel Servet (Other)
Other Study IDs: ALB-RME-2013-01
Record Dates: First submitted 2017-02-03; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Endoscopic Resection; Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational, prospective, multicentre and international study. This will be a non-interventional study to evaluate the efficacy and safety of endoscopic resection of gastrointestinal lesions and to determine what are the factors related to complications, and to describe these lesions according to the different morphologic and histologic classifications.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who are at least 18 years old.
* Clinical indication for endoscopic exam and endoscopic resection
* Patients must freely accept their involvement in this study. They shall give a written informed consent

Exclusion Criteria:

* Patients who do not desire to be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical indication for endoscopic resection at the different participating centers will be consecutively included in this study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-04-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of complete resections without recurrence | 6 month post-endoscopic resection

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Albeniz Arbizu, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Albeniz E, Gimeno-Garcia AZ, Fraile M, Ibanez B, Guarner-Argente C, Alonso-Aguirre P, Alvarez MA, Gargallo CJ, Pellise M, Ramos Zabala F, Herreros de Tejada A, Nogales O, Martinez-Ares D, Mugica F, de la Pena J, Espinos J, Huerta A, Alvarez A, Gonzalez-Santiago JM, Navajas F, Martinez-Cara JG, Redondo-Cerezo E, Merlo Mas J, Sabado F, Rivero L, Saperas E, Soto S, Rodriguez-Sanchez J, Lopez-Roses L, Rodriguez-Tellez M, Rullan Iriarte M, Elosua Gonzalez A, Pardeiro R, Valdivielso Cortazar E, Concepcion-Martin M, Huelin Alvarez P, Colan Hernandez J, Cobian J, Santiago J, Jimenez A, Remedios D, Lopez-Viedma B, Garcia O, Martinez-Alcala F, Perez-Roldan F, Carbo J, Enguita M. Clinical validation of risk scoring systems to predict risk of delayed bleeding after EMR of large colorectal lesions. Gastrointest Endosc. 2020 Apr;91(4):868-878.e3. doi: 10.1016/j.gie.2019.10.013. Epub 2019 Oct 23. PMID 31655045
- See also: Related Info — http://navarrabiomed.es